CLINICAL TRIAL: NCT04138654
Title: Natural Compounds to Reduce Nitrite in Meat Products: PHYTOME
Brief Title: Natural Compounds to Reduce Nitrite in Meat Products
Acronym: PHYTOME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL43956.068.13
Record Dates: First submitted 2014-01-08; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2014-01

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Poultry

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal nitrite levels (Experimental): Processed meat products enriched with natural compounds will contain normal nitrite levels.
  Interventions: Dietary Supplement: Processed meat product; Dietary Supplement: White meat wash-out; Dietary Supplement: Processed meat products enriched with natural compounds; Dietary Supplement: Drinking water containing nitrate up to acceptable daily intake level (ADI = 3.7 mg/kg bw) in combination with 300 grams of processed meat, white meat or processed meat enriched with natural compounds
- Reduced nitrite levels (Experimental): Processed meat products enriched with natural compounds will contain reduced nitrite levels
  Interventions: Dietary Supplement: Processed meat product; Dietary Supplement: White meat wash-out; Dietary Supplement: Processed meat products enriched with natural compounds; Dietary Supplement: Drinking water containing nitrate up to acceptable daily intake level (ADI = 3.7 mg/kg bw) in combination with 300 grams of processed meat, white meat or processed meat enriched with natural compounds

INTERVENTIONS:
Dietary Supplement: Processed meat product — 300 grams per day during 2 weeks
Dietary Supplement: White meat wash-out — 300 grams per day during 2 weeks
Dietary Supplement: Processed meat products enriched with natural compounds — 300 grams per day during 2 weeks
Dietary Supplement: Drinking water containing nitrate up to acceptable daily intake level (ADI = 3.7 mg/kg bw) in combination with 300 grams of processed meat, white meat or processed meat enriched with natural compounds — 3.7 mg nitrate/kg bw per day plus 300 grams of meat for 1 week

SUMMARY:
The PHYTOME project (Phytochemicals to reduce nitrite in meat products) is a major European Union (EU) co-funded research project that aims to develop innovative meat products in which the food additive nitrite has been replaced by natural compounds originating from fruits and vegetables. These biologically active compounds, also referred to as phytochemicals, are known to contribute to improved gut health and are added to the meat as natural extracts.

In a number of meat products, carefully selected combinations of natural antioxidants and other biologically active compounds occurring in vegetables, fruits and natural extracts such as coffee and tea, will be added during meat processing. Some of these compounds possess an antimicrobial activity allowing them to replace nitrite, whereas others possess a natural red colour that may contribute to the desired appearance of the products. Also, some of these compounds are known to protect colonic cells against damaging effects of cancer causing agents that may be formed in the large intestine after meat consumption.

The PHYTOME project will develop new technologies to introduce the natural extracts during processing to different types of meat products. These techniques will guarantee good sensory quality of the product as well as microbiological safety. Once these techniques have been developed and optimized at laboratory scale, the new type of products will be produced on an industrial scale. The health promoting effects of these products will be evaluated in a human dietary intervention study with healthy volunteers. After consumption of a fully controlled diet with either relatively high amounts of the traditional meat products or products produced following the new concept, faeces and colonic material will be collected and investigated for markers of colorectal cancer risk. These investigations will be performed in close collaboration with Research Institutes in the United Kingdom, Belgium, Italy and Greece, and will make use of the newest genomics techniques that are available.

DETAILED DESCRIPTION:
Rationale:

The aim of this project is to develop new meat processing technologies, resulting in innovative meat products that have low or no nitrite and that have been shown to contribute to improved human health. This will be achieved by introducing carefully selected mixtures of biologically compounds originating from natural plant extracts. The new meat products will be evaluated in a human dietary intervention study to establish their positive effect on cancer risk markers in colonic tissues using the newest genomics techniques available.

Objective:

This project aims to evaluate the health impact of newly developed low nitrite containing meat products using genomics markers in a human dietary intervention study.

Study design:

This study has a cross-over design with only healthy volunteers. Each participant will be asked to donate a urinal, faecal and blood sample and undergo endoscopy after each intervention period. All analyses will be done for each study group separately to examine the overall effects of nitrite levels in meat.

Study population:

All subjects will be recruited by the University of Maastricht (UM) in the province of Limburg, the Netherlands, using advertisements in local newspapers as well as other media. Healthy subjects of both sexes will be selected based on predefined inclusion criteria (BMI: 18-25; > 18 years) and randomly assigned to one of the different experimental groups.

Intervention (if applicable):

Subjects will receive a completely controlled diet with 3 different types of meat products according to the study design, with either normal levels, low or no added nitrite. After each of the three intervention periods of 15 days (300 grams meat per day) blood, urine, saliva, mouth wash and faeces will be sampled and stored appropriately at UM for later analysis. Additionally, colonic biopsies will be taken by the department of internal medicine (UM) or at the hospital of Sittard during an endoscopic examination. To evaluate the impact of nitrate in drinking water on the endogenous nitrosation processes in combination with processed red meat intake, there will be and extra intervention period of 7 days were volunteers will be asked to consume drinking water with high nitrate levels according to the Acceptable Daily Intake level (ADI: 3.7mg/kg bodyweight) in combination with 300 grams processed red meat per day. Also after this intervention period volunteers will be asked to collect a blood and saliva sample and 24h urine and faeces samples. Also, colonic biopsies will be taken by the department of internal medicine (UM) or at the hospital of Sittard during an endoscopic examination.

Main study parameters/endpoints:

* Formation of N-nitrosocompounds in human faecal and urine samples
* Reveal differences in transcriptomic and epigenomic markers after consumption of meat products enriched with natural compounds. These markers can be interpreted as an indicator of reduced cancer risk.
* Correlating gene expression changes to changes in genotoxic endpoints (DNA damage, reduction in N-Nitroso compounds (NOC)) to reveal the molecular processes involved in cancer risk reduction. The identification of molecular pathways that are crucial in the carcinogenic process will demonstrate a causal association between dietary changes and markers of carcinogenic risk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with a Body Mass Index (BMI) between 18-25, male or female
* Between 18-70 years old

Exclusion Criteria:

* Alcohol abuse up to 6 months before participation in this research
* Current aberrations or insufficiency of kidney, liver, gut, heart or lungs
* Current presence of persistent inflammation in the gut or liver
* Current endocrine or metabolic aberrations
* Current anaemia or infection
* HIV infection or hepatitis
* Use of antibiotics and other medication over the last 3 months
* Current smokers
* Vegetarians
* Pregnant women
* Participants of other intervention studies during this intervention period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Change in N-nitroso compound (NOC) levels in faeces and urine measured as apparent total nitroso compounds (ATNC) between baseline levels at the start of the intervention and each intervention period | At baseline, at 2 weeks, at 4 weeks, at 6 weeks, and at 7 weeks
  The faecal and urinal level of NOC is measured as Total Apparent Nitroso Compounds (ATNC) and used indicator of colonic endogenous nitrosation. It is known to significantly increase following strictly controlled diets high in red or processed meat.
Change in whole genome gene expression analyses in colonic biopsies and blood between baseline levels and each intervention period (transcriptomics) | At baseline, at 2 weeks, at 4 weeks, and at 6 weeks
  Colon biopsies and blood will be analysed for transcriptomic responses to the dietary changes. This will provide information on gene expression changes in the colon epithelium that may be linked with other parameters such as faecal NOC levels. This will also identify molecular pathways that can link dietary composition to processes involved in cancer development.

SECONDARY OUTCOMES:
Change in urinary nitrate and creatine levels between baseline levels at the start of the intervention and each intervention period. | At baseline, at 2 weeks, at 4 weeks, at 6 weeks, and at 7 weeks
  Urine samples (0.25 mL) will be analysed for nitrate and urinary creatinine. Nitrate concentrations (ng/ml) will be divided by creatinine concentrations (mg/100ml) to adjust for the variable hydration of participants.
Genotyping of DNA | At baseline
  Blood will be collected which will be used for genotyping of single nucleotide polymorphisms associated with oxidative stress, biotransformation and DNA repair. This will provide information on the relation between genetic variations linked with other tested parameters such as faecal NOC levels.
Change in DNA methylation analyses of DNA isolated from colonic biopsies and blood (epigenetics) between baseline levels at the start of the intervention and each intervention period | At baseline, at 2 weeks, at 4 weeks, at 6 weeks
  Colon biopsies and blood will be analysed for epigenomic responses to the dietary changes. This will provide information on the genes of which the DNA methylation status has changed which might explain their change in gene expression. Epigenetic changes and gene expression changes will be integrated during the analyses.
Change in enzyme activity of nitrate reductase in saliva between baseline levels at the start of the intervention and each intervention period | At baseline, at 2 weeks, at 4 weeks, at 6 weeks, and at 7 weeks
  Microorganisms in the mouth are able to convert nitrate to nitrite and it has been estimated that about 70% of ingested nitrite is formed in this way. Dietary interventions containing nitrate have shown to infuence the activity of the enzyme nitrate reductase.
Change in the microbiome in feacal samples and in saliva between baseline levels at the start of the intervention and each intervention period | At baseline, at 2 weeks, at 4 weeks, at 6 weeks, and at 7 weeks
  Both saliva and fecal specimens will be used for DNA extraction and subsequent analyses. The microbiome is sensitive for dietary changes, and its composition can alter due to different exposures.

OTHER OUTCOMES:
Change in faecal water genotoxicity between baseline levels at the start of the intervention and each intervention period | At baseline, at 2 weeks, at 4 weeks, at 6 weeks
  Faecal water can be prepared from faecal matter after which a short-term exposure of an in vitro colon cell line will be performed. DNA damage will subsequently be assessed by the alkaline single cell gel electrophoresis assay or comet assay.
Change in O6-CMG in colonic biopsies between baseline levels at the start of the intervention and each intervention period | At baseline, at 2 weeks, at 4 weeks, at 6 weeks
  O6-CMG is a mutagenic DNA adduct that results from exposure to nitrosated glycine derivatives and has particular potential as a biological marker of DNA carboxymethylation because it does not seem to be repaired by O6-alkylguaninealkyltransferase. O6-CMG has previously been found to increase following a diet high in red meat.
Change in O6-MeG in colonic biopsies between baseline levels at the start of the intervention and each intervention period | At baseline, at 2 weeks, at 4 weeks, at 6 weeks
  Exposure to certain NOCs causes O6-MeG adduct formation. O6-MeG DNA adducts are also mutagenic and have frequently been shown to occur in human CRC tissue. Samples will be analyzed at National Hellenic Research Foundation (NHRF; Greece) using an ELISA method described by Georgiadis et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Toxicogenomics, Maastricht, (Click to Select US State), Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Oliveira CE, Stamford TL, Gomes Neto NJ, de Souza EL. Inhibition of Staphylococcus aureus in broth and meat broth using synergies of phenolics and organic acids. Int J Food Microbiol. 2010 Feb 28;137(2-3):312-6. doi: 10.1016/j.ijfoodmicro.2009.11.019. Epub 2009 Dec 3. PMID 20004993
- [Background] Burt S. Essential oils: their antibacterial properties and potential applications in foods--a review. Int J Food Microbiol. 2004 Aug 1;94(3):223-53. doi: 10.1016/j.ijfoodmicro.2004.03.022. PMID 15246235
- [Background] Cheng KW, Chen F, Wang M. Inhibitory activities of dietary phenolic compounds on heterocyclic amine formation in both chemical model system and beef patties. Mol Nutr Food Res. 2007 Aug;51(8):969-76. doi: 10.1002/mnfr.200700032. PMID 17628877
- [Background] Hughes R, Cross AJ, Pollock JR, Bingham S. Dose-dependent effect of dietary meat on endogenous colonic N-nitrosation. Carcinogenesis. 2001 Jan;22(1):199-202. doi: 10.1093/carcin/22.1.199. PMID 11159760
- [Background] Lunn JC, Kuhnle G, Mai V, Frankenfeld C, Shuker DE, Glen RC, Goodman JM, Pollock JR, Bingham SA. The effect of haem in red and processed meat on the endogenous formation of N-nitroso compounds in the upper gastrointestinal tract. Carcinogenesis. 2007 Mar;28(3):685-90. doi: 10.1093/carcin/bgl192. Epub 2006 Oct 19. PMID 17052997
- [Background] Cross AJ, Major JM, Sinha R. Urinary biomarkers of meat consumption. Cancer Epidemiol Biomarkers Prev. 2011 Jun;20(6):1107-11. doi: 10.1158/1055-9965.EPI-11-0048. Epub 2011 Apr 28. PMID 21527577
- [Background] Hall CN, Badawi AF, O'Connor PJ, Saffhill R. The detection of alkylation damage in the DNA of human gastrointestinal tissues. Br J Cancer. 1991 Jul;64(1):59-63. doi: 10.1038/bjc.1991.239. PMID 1854628
- [Background] Povey AC, Badawi AF, Cooper DP, Hall CN, Harrison KL, Jackson PE, Lees NP, O'Connor PJ, Margison GP. DNA alkylation and repair in the large bowel: animal and human studies. J Nutr. 2002 Nov;132(11 Suppl):3518S-3521S. doi: 10.1093/jn/132.11.3518S. PMID 12421880
- [Background] Georgiadis P, Kaila S, Makedonopoulou P, Fthenou E, Chatzi L, Pletsa V, Kyrtopoulos SA. Development and validation of a new, sensitive immunochemical assay for O(6)-methylguanine in DNA and its application in a population study. Cancer Epidemiol Biomarkers Prev. 2011 Jan;20(1):82-90. doi: 10.1158/1055-9965.EPI-10-0788. Epub 2010 Nov 16. PMID 21081711
- [Background] MAQC Consortium; Shi L, Reid LH, Jones WD, Shippy R, Warrington JA, Baker SC, Collins PJ, de Longueville F, Kawasaki ES, Lee KY, Luo Y, Sun YA, Willey JC, Setterquist RA, Fischer GM, Tong W, Dragan YP, Dix DJ, Frueh FW, Goodsaid FM, Herman D, Jensen RV, Johnson CD, Lobenhofer EK, Puri RK, Schrf U, Thierry-Mieg J, Wang C, Wilson M, Wolber PK, Zhang L, Amur S, Bao W, Barbacioru CC, Lucas AB, Bertholet V, Boysen C, Bromley B, Brown D, Brunner A, Canales R, Cao XM, Cebula TA, Chen JJ, Cheng J, Chu TM, Chudin E, Corson J, Corton JC, Croner LJ, Davies C, Davison TS, Delenstarr G, Deng X, Dorris D, Eklund AC, Fan XH, Fang H, Fulmer-Smentek S, Fuscoe JC, Gallagher K, Ge W, Guo L, Guo X, Hager J, Haje PK, Han J, Han T, Harbottle HC, Harris SC, Hatchwell E, Hauser CA, Hester S, Hong H, Hurban P, Jackson SA, Ji H, Knight CR, Kuo WP, LeClerc JE, Levy S, Li QZ, Liu C, Liu Y, Lombardi MJ, Ma Y, Magnuson SR, Maqsodi B, McDaniel T, Mei N, Myklebost O, Ning B, Novoradovskaya N, Orr MS, Osborn TW, Papallo A, Patterson TA, Perkins RG, Peters EH, Peterson R, Philips KL, Pine PS, Pusztai L, Qian F, Ren H, Rosen M, Rosenzweig BA, Samaha RR, Schena M, Schroth GP, Shchegrova S, Smith DD, Staedtler F, Su Z, Sun H, Szallasi Z, Tezak Z, Thierry-Mieg D, Thompson KL, Tikhonova I, Turpaz Y, Vallanat B, Van C, Walker SJ, Wang SJ, Wang Y, Wolfinger R, Wong A, Wu J, Xiao C, Xie Q, Xu J, Yang W, Zhang L, Zhong S, Zong Y, Slikker W Jr. The MicroArray Quality Control (MAQC) project shows inter- and intraplatform reproducibility of gene expression measurements. Nat Biotechnol. 2006 Sep;24(9):1151-61. doi: 10.1038/nbt1239. PMID 16964229
- [Background] Jetten MJ, Gaj S, Ruiz-Aracama A, de Kok TM, van Delft JH, Lommen A, van Someren EP, Jennen DG, Claessen SM, Peijnenburg AA, Stierum RH, Kleinjans JC. 'Omics analysis of low dose acetaminophen intake demonstrates novel response pathways in humans. Toxicol Appl Pharmacol. 2012 Mar 15;259(3):320-8. doi: 10.1016/j.taap.2012.01.009. Epub 2012 Jan 20. PMID 22285215
- [Background] Mathijs K, Brauers KJ, Jennen DG, Boorsma A, van Herwijnen MH, Gottschalk RW, Kleinjans JC, van Delft JH. Discrimination for genotoxic and nongenotoxic carcinogens by gene expression profiling in primary mouse hepatocytes improves with exposure time. Toxicol Sci. 2009 Dec;112(2):374-84. doi: 10.1093/toxsci/kfp229. Epub 2009 Sep 21. PMID 19770486
- [Background] Mathijs K, Brauers KJ, Jennen DG, Lizarraga D, Kleinjans JC, van Delft JH. Gene expression profiling in primary mouse hepatocytes discriminates true from false-positive genotoxic compounds. Mutagenesis. 2010 Nov;25(6):561-8. doi: 10.1093/mutage/geq040. Epub 2010 Jul 21. PMID 20650930
- [Background] Tannenbaum SR, Sinskey AJ, Weisman M, Bishop W. Nitrite in human saliva. Its possible relationship to nitrosamine formation. J Natl Cancer Inst. 1974 Jul;53(1):79-84. No abstract available. PMID 4835100
- [Background] Shechter H, Gruener N, Shuval HI. A micromethod for the determination of nitrite in blood. Anal Chim Acta. 1972 Jun;60(1):93-9. doi: 10.1016/S0003-2670(01)81887-0. No abstract available. PMID 4667452
- [Result] Hodgson JM, Burke V, Beilin LJ, Puddey IB. Partial substitution of carbohydrate intake with protein intake from lean red meat lowers blood pressure in hypertensive persons. Am J Clin Nutr. 2006 Apr;83(4):780-7. doi: 10.1093/ajcn/83.4.780. PMID 16600928
- [Result] Bingham SA, Pignatelli B, Pollock JR, Ellul A, Malaveille C, Gross G, Runswick S, Cummings JH, O'Neill IK. Does increased endogenous formation of N-nitroso compounds in the human colon explain the association between red meat and colon cancer? Carcinogenesis. 1996 Mar;17(3):515-23. doi: 10.1093/carcin/17.3.515. PMID 8631138
- [Result] Cross AJ, Sinha R. Meat-related mutagens/carcinogens in the etiology of colorectal cancer. Environ Mol Mutagen. 2004;44(1):44-55. doi: 10.1002/em.20030. PMID 15199546
- [Result] Wakabayashi K, Nagao M, Esumi H, Sugimura T. Food-derived mutagens and carcinogens. Cancer Res. 1992 Apr 1;52(7 Suppl):2092s-2098s. PMID 1544146
- [Result] Kuhnle GG, Bingham SA. Dietary meat, endogenous nitrosation and colorectal cancer. Biochem Soc Trans. 2007 Nov;35(Pt 5):1355-7. doi: 10.1042/BST0351355. PMID 17956350
- [Result] Cross AJ, Pollock JR, Bingham SA. Haem, not protein or inorganic iron, is responsible for endogenous intestinal N-nitrosation arising from red meat. Cancer Res. 2003 May 15;63(10):2358-60. PMID 12750250
- [Result] Haorah J, Zhou L, Wang X, Xu G, Mirvish SS. Determination of total N-nitroso compounds and their precursors in frankfurters, fresh meat, dried salted fish, sauces, tobacco, and tobacco smoke particulates. J Agric Food Chem. 2001 Dec;49(12):6068-78. doi: 10.1021/jf010602h. PMID 11743810
- [Result] Ozel MZ, Gogus F, Yagci S, Hamilton JF, Lewis AC. Determination of volatile nitrosamines in various meat products using comprehensive gas chromatography-nitrogen chemiluminescence detection. Food Chem Toxicol. 2010 Nov;48(11):3268-73. doi: 10.1016/j.fct.2010.08.036. Epub 2010 Sep 8. PMID 20816717
- [Result] Hebels DG, Briede JJ, Khampang R, Kleinjans JC, de Kok TM. Radical mechanisms in nitrosamine- and nitrosamide-induced whole-genome gene expression modulations in Caco-2 cells. Toxicol Sci. 2010 Jul;116(1):194-205. doi: 10.1093/toxsci/kfq121. Epub 2010 Apr 19. PMID 20403970
- [Result] Hebels DG, Jennen DG, van Herwijnen MH, Moonen EJ, Pedersen M, Knudsen LE, Kleinjans JC, de Kok TM. Whole-genome gene expression modifications associated with nitrosamine exposure and micronucleus frequency in human blood cells. Mutagenesis. 2011 Nov;26(6):753-61. doi: 10.1093/mutage/ger043. Epub 2011 Jul 1. PMID 21724973
- [Result] Hebels DG, Sveje KM, de Kok MC, van Herwijnen MH, Kuhnle GG, Engels LG, Vleugels-Simon CB, Mares WG, Pierik M, Masclee AA, Kleinjans JC, de Kok TM. N-nitroso compound exposure-associated transcriptomic profiles are indicative of an increased risk for colorectal cancer. Cancer Lett. 2011 Oct 1;309(1):1-10. doi: 10.1016/j.canlet.2011.05.007. Epub 2011 Jun 12. PMID 21669488
- [Result] Hebels DG, Sveje KM, de Kok MC, van Herwijnen MH, Kuhnle GG, Engels LG, Vleugels-Simon CB, Mares WG, Pierik M, Masclee AA, Kleinjans JC, de Kok TM. Red meat intake-induced increases in fecal water genotoxicity correlate with pro-carcinogenic gene expression changes in the human colon. Food Chem Toxicol. 2012 Feb;50(2):95-103. doi: 10.1016/j.fct.2011.10.038. Epub 2011 Oct 14. PMID 22019696
- [Result] Honikel KO. The use and control of nitrate and nitrite for the processing of meat products. Meat Sci. 2008 Jan;78(1-2):68-76. doi: 10.1016/j.meatsci.2007.05.030. Epub 2007 Jun 27. PMID 22062097
- [Result] Lee SY, Munerol B, Pollard S, Youdim KA, Pannala AS, Kuhnle GG, Debnam ES, Rice-Evans C, Spencer JP. The reaction of flavanols with nitrous acid protects against N-nitrosamine formation and leads to the formation of nitroso derivatives which inhibit cancer cell growth. Free Radic Biol Med. 2006 Jan 15;40(2):323-34. doi: 10.1016/j.freeradbiomed.2005.08.031. Epub 2005 Oct 11. PMID 16413414
- [Result] Pollard SE, Kuhnle GG, Vauzour D, Vafeiadou K, Tzounis X, Whiteman M, Rice-Evans C, Spencer JP. The reaction of flavonoid metabolites with peroxynitrite. Biochem Biophys Res Commun. 2006 Dec 1;350(4):960-8. doi: 10.1016/j.bbrc.2006.09.131. Epub 2006 Oct 2. PMID 17045238
- [Result] de Kok TM, van Breda SG, Manson MM. Mechanisms of combined action of different chemopreventive dietary compounds: a review. Eur J Nutr. 2008 May;47 Suppl 2:51-9. doi: 10.1007/s00394-008-2006-y. PMID 18458834
- [Result] Bartsch H, Frank N. Blocking the endogenous formation of N-nitroso compounds and related carcinogens. IARC Sci Publ. 1996;(139):189-201. PMID 8923031
- [Result] Ward MH, Heineman EF, Markin RS, Weisenburger DD. Adenocarcinoma of the stomach and esophagus and drinking water and dietary sources of nitrate and nitrite. Int J Occup Environ Health. 2008 Jul-Sep;14(3):193-7. doi: 10.1179/oeh.2008.14.3.193. PMID 18686719
- [Result] Rowland IR, Granli T, Bockman OC, Key PE, Massey RC. Endogenous N-nitrosation in man assessed by measurement of apparent total N-nitroso compounds in faeces. Carcinogenesis. 1991 Aug;12(8):1395-401. doi: 10.1093/carcin/12.8.1395. PMID 1860160
- [Result] Kuhnle GG, Story GW, Reda T, Mani AR, Moore KP, Lunn JC, Bingham SA. Diet-induced endogenous formation of nitroso compounds in the GI tract. Free Radic Biol Med. 2007 Oct 1;43(7):1040-7. doi: 10.1016/j.freeradbiomed.2007.03.011. Epub 2007 Mar 13. PMID 17761300
- [Result] Lewin MH, Bailey N, Bandaletova T, Bowman R, Cross AJ, Pollock J, Shuker DE, Bingham SA. Red meat enhances the colonic formation of the DNA adduct O6-carboxymethyl guanine: implications for colorectal cancer risk. Cancer Res. 2006 Feb 1;66(3):1859-65. doi: 10.1158/0008-5472.CAN-05-2237. PMID 16452248
- [Result] Kok TM, Breda SG, Briede JJ. Genomics-based identification of molecular mechanisms behind the cancer preventive action of phytochemicals: potential and challenges. Curr Pharm Biotechnol. 2012 Jan;13(1):255-64. doi: 10.2174/138920112798868601. PMID 21466423
- [Derived] Sinha R, Zhao N, Goedert JJ, Byrd DA, Wan Y, Hua X, Hullings AG, Knight R, Breda SV, Mathijs K, de Kok TM, Ward MH; PHYTOME consortium members. Effects of processed meat and drinking water nitrate on oral and fecal microbial populations in a controlled feeding study. Environ Res. 2021 Jun;197:111084. doi: 10.1016/j.envres.2021.111084. Epub 2021 Mar 27. PMID 33785324